CLINICAL TRIAL: NCT02854514
Title: Predictive Value of Endometrial Cytokines in Endometrial Implantation in Cases of Intracytoplasmic Sperm Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, director clinical research, Benha University
Other Study IDs: Khalid 2
Record Dates: First submitted 2016-07-30; First posted 2016-08-03 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
Keywords: endometrial -cytokines
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aspiration of endometrial secretion: intra uterine flushing of the endometrial cavity by five millilitre of saline through embryo transfer catheter then aspirated with endometrial secretion then centrifuged then analyzed for detection of concentration of tumor necrosis factor a and interleukin 1 b
  Interventions: Procedure: Aspiration of endometrial secretion

INTERVENTIONS:
Procedure: Aspiration of endometrial secretion — intra uterine flushing of the endometrial cavity by five millilitre of saline through embryo transfer catheter then aspirated then centrifuged then analyzed for detection of concentration of tumor necrosis factor a and interleukin 1 b

SUMMARY:
For all women immediately after ovum retrieval from 80 women undergoing IVF, intra uterine salin flushing will be analyzed using a multiplex immunoassay for soluble regulators of implantation, namely Interleukin (IL)-1b, Tumor Necrosis Factor (TNF)-a,. In order to detect implantation predictors.

DETAILED DESCRIPTION:
This is a prospective cohort study, performed on 80 women attending Obstetrics and Gynecology Department of Benha University Hospital for invitro fertilization/intracytoplasmic sperm injection treatment and private IVF centers. None undergoes more than one prior unsuccessful embryo transfer.

Method of randomization:

Simple random sample, which is a subset of individuals (a sample) chosen from a larger set (a population). Each individual is chosen randomly and entirely by chance, so each individual has the sample probability of being chosen at any stage during the sampling process, and each subset of k individuals has the same probability of being chosen for the sample as any other subset of k individuals (Yates et al., 2008).

Methods:

The patients will be subjected to the following:

* History.
* General examination.
* Endometrial secretion aspiration.
* Determination of the cytokine profile.
* Detection of implantation rate.

Inclusion criteria:

1. Age younger than 37 years.
2. Having a regular and proven ovulatory menstrual cycles with a length of 26-35 days.
3. Body mass index less than 35 kg/m2.
4. Serum follicle stimulating hormone and estradiol were within normal ranges.

Indications of IVF:

Tubal pathology, unexplained infertility, and male factor.

Exclusion criteria:

Gross uterine pathology.

Steps of performance:

All women having the inclusion criteria were subjected to super ovulation protocols followed by hcg adminstration when the follicles reached 18-20 mm . Ovum retrieval were done at 35 hours following hcg injection.

Five millilitre of salin are injected intrauterine then aspirated after ovum retrieval.Endometrial secretions, aspirated immediately after ovum retrieval from 80 women undergoing IVF, will be analyzed using a multiplex immunoassay for soluble regulators of implantation, namely Interleukin (IL)-1b, Tumor Necrosis Factor (TNF)-a,. In order to detect implantation predictors.

ELIGIBILITY:
Inclusion Criteria:

1. Age younger than 37 years.
2. Having a regular and proven ovulatory menstrual cycles with a length of 26-35 days.
3. Body mass index less than 35 kg/m2.
4. Serum follicle stimulating hormone and estradiol were within normal ranges.

Exclusion Criteria:

* Gross uterine pathology.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients undergoing IVF
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Tumor Necrosis Factor (TNF)-a | 2 days
Measurement of Interleukin (IL)-1b | 2 days

SECONDARY OUTCOMES:
serum pregnancy test | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: khalid M salama, MD, Study Director — Benha University
Locations (1):
- Benha university, Banhā, Al Qalubia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boomsma CM, Kavelaars A, Eijkemans MJ, Amarouchi K, Teklenburg G, Gutknecht D, Fauser BJ, Heijnen CJ, Macklon NS. Cytokine profiling in endometrial secretions: a non-invasive window on endometrial receptivity. Reprod Biomed Online. 2009 Jan;18(1):85-94. doi: 10.1016/s1472-6483(10)60429-4. PMID 19146774
- [Derived] Salama KM, Alloush MK, Al Hussini RM. Are the cytokines TNF alpha and IL 1Beta early predictors of embryo implantation? Cross sectional study. J Reprod Immunol. 2020 Feb;137:102618. doi: 10.1016/j.jri.2019.102618. Epub 2019 Oct 17. PMID 31698104